CLINICAL TRIAL: NCT05581173
Title: Multicenter Prospective Evaluation of the Efficacy of a Self-Assembling Matrix Forming Gel to Prevent Stricture Formation in High-Risk Patients
Brief Title: Self-Assembling Matrix Forming Gel to Prevent Stricture Formation
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1931151
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Stricture; Stricture
MeSH Terms: conditions — Esophageal Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic resection of gastrointestinal lesion(s): Endoscopic mucosal resection or endoscopic submucosal dissection is an outpatient procedure to remove superficial neoplasia(precancerous lesions and early cancer) throughout the gastrointestinal tract.
  Interventions: Device: Purastat SAP gel application

INTERVENTIONS:
Device: Purastat SAP gel application — Purastat is a fully synthetic matrix scaffold that can be applied through an endoscopic catheter. Purastat is FDA approved and commercially available. Purastat is a peptide solution that self assembles at physiological potential Hydrogen(pH) and forms a gel comprising a network of nanofibers. Its benefits in hemostasis and tissue healing and its biocompatibility have been previously demonstrated in animal models and also in human cases. When the gel comes into contact with blood or tissue fluids, the change in potential hydrogen (pH) and salt concentration causes fiber formation and gelation that block the blood vessels in the hemorrhagic area to generate hemostatic effects and also prevention of scar tissue formation.

SUMMARY:
The study is designed as a multicenter prospective registry study evaluating the efficacy of the self-assembling peptide in the prevention of stricture formation after endoscopic resection as part of standard medical care. No experimental interventions will be performed.

DETAILED DESCRIPTION:
In recent years, endoscopic resection by endoscopic mucosal resection(EMR) or endoscopic submucosal dissection(ESD) has become standard practice for the removal of superficial neoplasia (precancerous lesions and early cancer) throughout the gastrointestinal tract. These procedures are associated with lower morbidity and mortality when compared to conventional surgery.

Nonetheless, stricture formation following endoscopic resection of gastrointestinal lesions is a well-known risk, particularly in the esophagus. The main risk factor for esophageal stricture formation following EMR/ESD is resection size, with this increasing with the length and extent of the circumferential excision, reaching 100% stricture formation when the entire circumference is involved. Stricture formation is associated with significant morbidity and increasing health care utilization, as multiple endoscopies are often required as part of the management of these difficult to treat strictures.

Recently, a self-assembling peptide (SAP) forming gel (Purastat; 3D Matrix, Ltd, Tokyo, Japan) has been approved by the Food and Drug Administration (FDA) as an agent that that promotes healing, which may potentially reduce the risk of stricture formation. Initial small studies from Europe appear to show benefit but the magnitude of the effect has not been well defined. Furthermore, large prospective US based studies are currently lacking. Therefore, the aim of this study is to assess the efficacy of this novel SAP gel in the prevention of stricture formation after endoscopic resection in high-risk patients as utilized as part of clinically indicated standard patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients at high-risk for esophageal stricture formation defined as undergoing endoscopic resection in the esophagus involving more than 50% of the circumference

Exclusion Criteria:

* Any standard contraindication to anesthesia and/or endoscopy
* Participation in another research protocol that could interfere or influence the outcomes measures of the present study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to the participating centers for endoscopic resection of GI lesions may be eligible for entry into the study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Rate of stricture formation | 12 months
  Esophageal stricture will be defined as symptoms of dysphagia with concomitant endoscopy showing an inability to pass a standard endoscope due to luminal narrowing at the site of the resection scar.

SECONDARY OUTCOMES:
Workability of self-assembling peptide (SAP) gel application | 12 months
  The ability to adequately apply the SAP gel over the ulcer bed following resection.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — AdventHealth
Locations (6):
- United States (6):
  - AdventHealth Orlando, Orlando, Florida
  - Parkview, Fort Wayne, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Baylor St. Lukes, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gil ES, Aleksi E, Spirio L. PuraStat RADA16 Self-Assembling Peptide Reduces Postoperative Abdominal Adhesion Formation in a Rabbit Cecal Sidewall Injury Model. Front Bioeng Biotechnol. 2021 Dec 10;9:782224. doi: 10.3389/fbioe.2021.782224. eCollection 2021. PMID 34957076
- [Background] Subramaniam S, Kandiah K, Thayalasekaran S, Longcroft-Wheaton G, Bhandari P. Haemostasis and prevention of bleeding related to ER: The role of a novel self-assembling peptide. United European Gastroenterol J. 2019 Feb;7(1):155-162. doi: 10.1177/2050640618811504. Epub 2018 Nov 5. PMID 30788128
- [Background] Wong E, Ho J, Smith M, Sritharan N, Riffat F, Smith MC. Use of Purastat, a novel haemostatic matrix based on self-assembling peptides in the prevention of nasopharyngeal adhesion formation. Int J Surg Case Rep. 2020;70:227-229. doi: 10.1016/j.ijscr.2020.04.027. Epub 2020 May 8. PMID 32422584
- [Background] Yu M, Tan Y, Liu D. Strategies to prevent stricture after esophageal endoscopic submucosal dissection. Ann Transl Med. 2019 Jun;7(12):271. doi: 10.21037/atm.2019.05.45. PMID 31355238
- [Background] Uraoka T, Ochiai Y, Fujimoto A, Goto O, Kawahara Y, Kobayashi N, Kanai T, Matsuda S, Kitagawa Y, Yahagi N. A novel fully synthetic and self-assembled peptide solution for endoscopic submucosal dissection-induced ulcer in the stomach. Gastrointest Endosc. 2016 Jun;83(6):1259-64. doi: 10.1016/j.gie.2015.11.015. Epub 2015 Dec 1. PMID 26608126